CLINICAL TRIAL: NCT03340831
Title: Post Approval Study for Non-Adjunctive Use of Dexcom G5 and G6 CGM System for Diabetes Management
Brief Title: Continuous Monitoring and Control of Hypoglycemia
Acronym: COACH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-901895
Record Dates: First submitted 2017-10-31; First posted 2017-11-14 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CGM/BGM Group: single-group, whereby participant is their own control. Use of a Blood Glucose Meter (BGM) for 6 months is compared to use of the G5 and G6 CGM System for 6 months, with collection of major diabetes related events (mild/severe hypoglycemia and DKA).
  Interventions: Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) — Use of CGM to compare incidence of diabetes events compared to use of a blood glucose meter (BGM)

SUMMARY:
Evaluate safety of non-adjunctive CGM use in CGM naive participants.

DETAILED DESCRIPTION:
The study comprises recruitment and consenting of pediatric and adult participants. At entry, the following information will be collected: demographics, labs, clinical and diabetes history information (history of mild/severe hypoglycemia or DKA events in the past 6 months and SMBG testing frequency). There are 3 clinic visits: Study Entry, Month 6 and Month 12 . Monthly phone contacts will be made to assess for any mild/severe hypoglycemic or DKA events and any details surrounding an event. Clinic visits at Months 6 and 12 will capture frequency of SMBG testing, A1C level and PRO information. CGM data will be obtained during the study to assess for CGM adherence.

ELIGIBILITY:
Inclusion Criteria:

* Naïve to real-time CGM
* Type 1 or insulin-requiring Type 2 diabetes
* ≥ 2 years old

Exclusion Criteria:

* Use of RT-CGM, within the past 12 months
* Pregnancy
* Concomitant disease or condition that may compromise patient safety including and not limited to severe mental illness, a diagnosed or suspected eating disorder or any uncontrolled long term medical condition that would interfere with study related tasks or visits, or ongoing treatment for a significant malignancy.
* Known (or suspected) significant allergy to medical grade adhesives
* Dialysis

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and pediatrics (2 or older), naïve to CGM, with Type 1 or insulin-requiring Type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1388 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in hypoglycemic events | 6 months
  Change in average number of hypoglycemic events per patient between CGM use compared to BGM use

SECONDARY OUTCOMES:
Change in A1C | 6 months
  Percent change in A1C lab between CGM use period compared to BGM use period.
Change in incidence of hypoglycemic events | 6 months
  Percent change of participants with at least one event between CGM use period compared to BGM use period.
Change in GMSS PRO scores | 6 months
  Percent change in mean scores for the Glucose monitoring satisfaction survey (GMSS) [Emotional and Trust subscales] between CGM use period compared to BGM use period.
Change in Diabetes Distress Scale (DDS) PRO scores | 6 months
  Percent change in mean scores for the DDS between CGM use period compared to BGM use period.
Change in Hypoglycemia Fear PRO scores | 6 months
  Percent change in mean scores for the Hypoglycemia Fear Survey between CGM use period compared to BGM use period.
Change in Hypoglycemia Confidence PRO scores | 6 months
  Percent change in mean scores for the Hypoglycemia Confidence Scale between CGM use period compared to BGM use period.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Director — Dexcom-Medical Affairs
Locations (25):
- United States (25):
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Diabetes and Endocrine Associates, La Mesa, California
  - Centre of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Mills-Peninsula Medical Center, San Mateo, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Florida Pediatric Endocrinology, Gainesville, Florida
  - Intervent Clinical Research Center, Pembroke Pines, Florida
  - University of South Florida Clinical Research Center, Tampa, Florida
  - Atlanta Diabetes, Atlanta, Georgia
  - Rocky Mountain Diabetes Center, Idaho Falls, Idaho
  - Northshore University Health System, Skokie, Illinois
  - Iowa Diabetes & Endocrinology Research Center, Des Moines, Iowa
  - Cotton O'Neil Clinical Research, Topeka, Kansas
  - International Diabetes Research Center, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Methodist Physicians Clinic - Diabetes and Endocrine Specialists, Omaha, Nebraska
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - University of Oklahoma Health Sciences Center Department of Pediatric Diabetes and Endocrinology, Oklahoma City, Oklahoma
  - Vanderbilt Eskind Diabetes Clinic, Nashville, Tennessee
  - Amarillo Medical Specialists, LLP, Amarillo, Texas
  - Texas Diabetes and Endocrine, Austin, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Advanced Research Associates, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No